CLINICAL TRIAL: NCT01861561
Title: Efficacy and Infectious Complications of Induction Therapy With Low-dose Versus High-dose Intravenous Cyclophosphamide for Proliferative Lupus Nephritis in Children
Brief Title: Low-dose VS High-dose IV Cyclophosphamide for Proliferative LN in Children
Acronym: Low/highIVCY
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The duration of the study is longer than 5 years and we can not recruit the participants to the target number.
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 125/2556(EC2)
Record Dates: First submitted 2013-05-19; First posted 2013-05-23 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Renal Insufficiency; Infection
MeSH Terms: conditions — Renal Insufficiency; Infections | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-dose intravenous cyclophosphamide (Experimental): Low-dose intravenous cyclophosphamide 500 mg/m2/dose every 4 weeks/months for 7 doses. Total duration is 6 months for the induction treatment.
  Interventions: Drug: Low-dose intravenous cyclophosphamide
- High-dose intravenous cyclophosphamide (Active Comparator): High-dose intravenous cyclophosphamide 1,000 mg/m2/dose, the first dose will be started with 500 mg/m2/dose and steped up to 750 mg/m2/dose for the second dose. Then the dosage will be increased to 1,000 mg/m2/dose for the third dose and continued the dosage through the seventh dose. Total duration is 6 months for the induction treatment.
  Interventions: Drug: High-dose intravenous cyclophosphamide

INTERVENTIONS:
Drug: Low-dose intravenous cyclophosphamide — Intravenous cyclophosphamide 500 mg/m2/dose every 4 weeks/months, total 7 doses
  Other Names: Cytoxan
  Arms: Low-dose intravenous cyclophosphamide
Drug: High-dose intravenous cyclophosphamide — Intravenous cyclophosphamide every 4 weeks/months, total in 7 doses:
  the 1st dose-500 mg/m2/dose,the 2nd dose-750 mg/m2/dose, the 3rd-7th doses- 1,000 mg/m2/dose with the maximum dose at 1,500 mg/dose
  Other Names: Cytoxan
  Arms: High-dose intravenous cyclophosphamide

SUMMARY:
Proliferative lupus nephritis (LN)is the predominant cause of morbidity and mortality in juvenile Systemic Lupus Erythematosus (SLE). Induction therapy with high-dose intravenous cyclophosphamide can improve renal outcomes, but considerably associated with infection. Although severe infection is the significant complication related to poorer prognosis for juvenile SLE patients in Asia, cyclophosphamide is still commonly used as the drug of choice for severe lupus nephritis. Euro-Lupus Nephritis Trial demonstrated low-dose intravenous cyclophosphamide regimen followed by azathioprine achieved good clinical results comparable with obtained high-dose regimen. There was lower number of severe infection episodes, but no significant difference. Recent studies applied low dose of cyclophosphamide (500 mg/m2/dose or 500 mg/dose)in young patients and showed good renal response. Low-dose intravenous cyclophosphamide regimen might promote non-inferior renal remission whereas decrease risk of serious infection and improve overall patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Child up to 15 years of age who fulfilled the 1997 updating the American College of Rheumatology revised criteria for the classification of SLE and his or her renal biopsy reveals lupus nephritis class III or IV regarding to International Society of Nephrology/Renal Pathology Society revision on the classification of the lupus nephritis.

Exclusion Criteria:

* patient who has prior renal insufficiency due to chronic kidney disease other than lupus nephritis
* patient who has the history of cyclophosphamide hypersensitivity
* patient who has prior cyclophosphamide or mycophenolate mofetil administration within 6 months
* patient who is pregnant

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2013-05; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
renal response | at 6 months of the treatment
  3 main renal parameters: renal function(eCCl),proteinuria(spot urine protein/creatinine ratio, UPCR), and urine sediment (rbc,wbc,and casts) 'renal remission'
  * complete- normal renal function, UPCR<0.2, and normal urine sediment(rbc<5,wbc<5/HPF,and no cast)
  * partial- at least 50%improvement in 2 main parameters with UPCR <= 1.0 and without worsening of remaining main parameter

SECONDARY OUTCOMES:
infection | within 6 months
  infectious episode classified in 3 levels
  * mild infection - the infection that is not serious and the patient could be treated with oral antimicrobial agent in outpatient clinic
  * moderate infection - the infection that the patient need admission or intravenous antimicrobial agent
  * serious infection - the infection that the patient is critically ill and need ICU care

OTHER OUTCOMES:
Patient well being | at 0,1,3 and 6 months of the treatment
  using visual analogue scale (VAS 0-10)for self assessment their well being
SLE disease activity index score | at 0,1,3 and 6 months of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nuntawan Piyaphanee, MD, Principal Investigator — Siriraj Hospital; Anirut Pattaragarn, MD, Study Director — Siriraj Hospital
Locations (1):
- Nephrology division, Department of Pediatrics, Siriraj Hospital, Bangkoknoi, Bangkok, Thailand